CLINICAL TRIAL: NCT07139769
Title: The RAISE Study: Adapting Psychosocial Resiliency Intervention for Parents of Adolescents and Young Adults With Cancer
Brief Title: Adapting Psychosocial Resiliency Intervention for Parents of Adolescents and Young Adults With Cancer
Acronym: RAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeba Ahmad, Ph.D. (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Zeba Ahmad, Ph.D., Clinical Staff Psychologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-242; IRG-21-130-10-IRG-11 (Other Grant/Funding Number: American Cancer Society Institutional Research Grant)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Caregiving for Cancer
Keywords: adolescents and young adults with cancer; cancer caregivers
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial Intervention for Parental Caregivers of AYA with Cancer (Experimental): The study team aims to evaluate the feasibility and acceptability of the adapted psychosocial intervention to 1) improve psychological resiliency to stress and 2) reduce symptoms of depression, anxiety, and post-traumatic stress among parental caregivers, through a single-arm open pilot trial of 32 parents.
  Interventions: Behavioral: Psychosocial Intervention for Parental Caregivers of AYA with Cancer

INTERVENTIONS:
Behavioral: Psychosocial Intervention for Parental Caregivers of AYA with Cancer — A new adaptation of an evidence-supported intervention, the SMART-3RP program, to address psychological symptoms and promote well-being among parental caregivers of AYA with cancer.

SUMMARY:
The study team aims to adapt a psychosocial intervention to reduce psychological distress among the caregiving parents of adolescents and young adults (aged 15-39) who have cancer. First, the study team will adapt an evidence-supported, group-based program for improving psychological resiliency (Stress Management and Resiliency Training - Relaxation Response Resiliency Program; SMART-3RP(E. R. Park et al., 2021)), and iteratively incorporate feedback from parents of AYA with cancer using a mixed-methods approach. Next, the study team will pilot the refined intervention to assess for preliminary indicators of feasibility, acceptability, and potential for efficacy in reducing parental distress.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying parent/guardian who provides a primary informal caregiving role in their child's cancer
* Recipient of caregiving is aged between 15 and 39 years and is receiving treatment for cancer
* Participant must score equal to or greater than 2 (out of a possible 10) on the National Comprehensive Cancer Network Distress Thermometer
* English-speaking
* Aged over 18 years

Exclusion Criteria:

* Having a co-parent or other household member participating in the same study
* Active symptoms of psychosis or suicidal ideation that would preclude safe participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility: Percent of Identified Prospective Participants Who Enroll | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Percent of eligible participants who were offered participation and who enroll in the study by completing consent and baseline assessment.
Intervention Feasibility: Proportion of Participants Completing the Program | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Percent of enrolled participants who complete the program, defined as completing 6 out of 8 sessions.
Intervention Acceptability | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Acceptability will be assessed by the Client Satisfaction Questionnaire (CSQ-8). The intervention study will be considered acceptable if ≥80% of participants rate it as acceptable (defined as a CSQ-8 score ≥20).

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham Cancer Institute at Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No